CLINICAL TRIAL: NCT02112448
Title: Continuous Infusion Versus Bolus Dosing for Pain Control After Pediatric Cardiothoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K5900208
Record Dates: First submitted 2014-03-28; First posted 2014-04-14 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-09

CONDITIONS: Congenital Heart Disease
Keywords: congenital heart disease, pediatric cardiothoracic surgery
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Acetaminophen; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous infusion (Active Comparator): Patients in this group will received morphine/midazolam drips at 0.3 mg/kg/hour each. They will be given doses of morphine 0.05 mg/kg/dose every 2 hours as needed for pain score 4 or more. Midazolam will also be given as needed (0.05 mg/kg/dose every 1 hour)
  Interventions: Drug: continuous infusion; Drug: Acetaminophen; Drug: ketorolac
- As needed dosing (Active Comparator): Patients in this arm will be given doses of morphine 0.05 mg/kg/dose every 2 hours as needed for pain score 4 or more. Midazolam will also be given as needed (0.05 mg/kg/dose every 1 hour)
  Interventions: Drug: as needed dosing; Drug: Acetaminophen; Drug: ketorolac

INTERVENTIONS:
Drug: continuous infusion — Continuous morphine/midazolam and 'as needed' doses. Will receive scheduled acetaminophen and ketorolac.
  Other Names: acetaminophen and ketorolac are scheduled for this arm of the study
  Arms: Continuous infusion
Drug: as needed dosing — morphine and midazolam as needed. Will receive scheduled acetaminophen and ketorolac..
  Other Names: acetaminophen and ketorolac are both scheduled for this arm as well
  Arms: As needed dosing
Drug: Acetaminophen — Acetaminophen will be given every 4 hours for a total of 24 hours.
Drug: ketorolac — Ketorolac 0.5 mg/kg will be given every six hours to all subjects in the study.

SUMMARY:
The investigators hypothesize that intermittent bolus doses of morphine and midazolam can provide the same pain control after pediatric cardiothoracic surgery as bolus doses plus infusions while using smaller total doses of both medications.

The investigators will randomize patients to receive either morphine/midazolam as needed intermittently or morphine/midazolam drips plus intermittent doses to be received as needed. Pain scores will be recorded and total medications given will be recorded.

DETAILED DESCRIPTION:
Prior to surgery, eligible patients scheduled for surgery will be sent our standard surgery letter (Attachment A) along with our study informational sheet (Attachment B) describing our study. The study informational sheet will have a telephone number to call to set up a phone appointment to discuss the study with the PI should parents have questions not answered on the sheet. During the pre-operative visit, the study will again be discussed with the parents. Our nurse practitioners will be trained on this study and will obtain written consent at this time. If the parents would like to further discuss the study directly with the PI, this will be arranged prior to surgery.

The PI will be notified by the NPs of all parents who give permission for their child to participate in the study, and he will notify the on service medical team. On the day of surgery, a computerized order for the study will be entered to notify the pharmacy to randomize the subject to the control or treatment group. Randomization will be stratified based on whether the child has DS, as children with DS are known to have a heightened pain response and require large doses of medication to treat pain. Only the pharmacist will know the random assignment, health care providers and subjects/families will be blinded as to treatment arm.

Treatment Group:

Intravenous (IV) drip of 0.03 mg/kg/hour morphine and 0.03 mg/kg/hour midazolam

Control Group:

IV drip of normal saline (NS) at same volume as what the morphine/midazolam drip would be

Both Groups

Subjects in both the control and treatment group will receive the following post-operative pain control orders that are currently in use in the PSHU:

1. Morphine 0.05 mg/kg/dose IV q 2 hours prn pain score 4 or greater
2. Midazolam 0.05 mg/kg/dose IV q1 hours prn agitation
3. Additional prn doses of morphine and midazolam may be given as determined by the treating team (these doses will be recorded in the EMR)
4. Acetaminophen 30 mg/kg PR x 1 to be given on admission to PSHU post surgery
5. Acetaminophen 15 mg/kg PR q4 hours to be started 4 hours after first dose
6. Acetaminophen 15 mg/kg PO q4 hours to be started after subject starts drinking by mouth and PR doses stopped
7. Ketorolac 0.5 mg/kg/dose IV q 6 hours to start 6-12 hours after surgery when chest tube drainage criteria are met. Will start when chest tube drainage is no longer frankly bloody and if chest tube drainage is less than 3 cc/kg/hour for two hours in a row

ELIGIBILITY:
Inclusion Criteria:

* Age 3 months - 4 years (48 months)
* Anticipated cardiothoracic surgery with midline sternotomy incision
* Planned early extubation (e.g. within 3 hours post surgery)

Exclusion Criteria:

* Presence of renal insufficiency defined as a creatinine greater than 0.8mg/dL on the standard basic metabolic profile sent after surgery or history of chronic renal failure.
* Significant development delay that the bedside nurse or treating physician judges would make pain scoring difficult (Down syndrome is not excluded)
* History of bleeding disorder or gastrointestinal bleed within the past 2 months.
* Presence of chronic hepatic disease or elevation of AST or ALT greater than 250 U/L before or after surgery.
* More than 3 previous surgeries with a sternotomy incision (this may alter pain perception).
* Children on immunosuppressants

Ages: 3 Months to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2014-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie S Penk, Principal Investigator — Advocate Children's Hospital
Locations (1):
- Advocate Children's Hospital, Oak Lawn, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled 78, but 18 were excluded after informed consent for the reasons listed below. 30 in each group were assigned and completed the study.
Groups:
- As Needed Dosing: Patients in this arm will be given doses of morphine 0.05 mg/kg/dose every 2 hours as needed for pain score 4 or more. Midazolam will also be given as needed (0.05 mg/kg/dose every 1 hour)
  as needed dosing: This group will receive morphine and midazolam as needed to control their pain. Acetaminophen and ketorolac will also be given for pain control in the same manner as the continuous infusion group.
  Acetaminophen: Acetaminophen will be given as a loading dose of 30 mg/kg rectally post surgery to all subjects and then 15 mg/kg every 4 hours for a total of 24 hours.
  ketorolac: Ketorolac 0.5 mg/kg will be given every six hours to all subjects in the study.
- Continuous Infusion: Patients in this group will received morphine/midazolam drips at 0.3 mg/kg/hour each. They will be given doses of morphine 0.05 mg/kg/dose every 2 hours as needed for pain score 4 or more. Midazolam will also be given as needed (0.05 mg/kg/dose every 1 hour)
  continuous infusion: This arm will receive continuous morphine/midazolam and 'as needed' doses. This group will receive adjunctive medications, acetaminophen and ketorolac.
  Acetaminophen: Acetaminophen will be given as a loading dose of 30 mg/kg rectally post surgery to all subjects and then 15 mg/kg every 4 hours for a total of 24 hours.
  ketorolac: Ketorolac 0.5 mg/kg will be given every six hours to all subjects in the study.
Period: Overall Study
Arm/Group | As Needed Dosing | Continuous Infusion
Started | 38 | 40
Completed | 30 | 30
Not Completed | 8 | 10
Not completed — lab values precluding use of ketorolac | 2 | 2
Not completed — Protocol Violation | 1 | 2
Not completed — Physician Decision | 4 | 6
Not completed — required heparin so could not use ketoro | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Infusion | As Needed Dosing | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: months] | 14.8 (12.1) | 16 (12.8) | 15.4 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 13 | 12 | 25
Presence of Down syndrome [Count of Participants; unit: Participants] | 5 | 4 | 9
Surgical complexity scores [Number; unit: units on a scale] — Surgical complexity scores are numbers assigned to a surgery type and range from 1-5 with 5 being the most complex. We added the surgical complexity scores of each patient and compared the sum between groups.
  units on a scale | 59 | 61 | 120

OUTCOME MEASURES:

1. Primary Outcome: Total Morphine Dosage
Description: Total dose of morphine used will be recorded for each patient.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Continuous Infusion | As Needed Dosing
Number analyzed (Participants) | 30 | 30
mg/kg | 0.9 (0.13) | 0.23 (0.14)

2. Secondary Outcome: Length of Stay
Description: Length of stay will be recorded for each subject.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause or discharge, whichever came first, assessed up to 100 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | As Needed Dosing | Continuous Infusion
Number analyzed (Participants) | 30 | 30
days | 4.9 (2.5) | 8.4 (7.7)

ADVERSE EVENTS:
Arm/Group | As Needed Dosing | Continuous Infusion
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/38 | 1/40
Other Adverse Events (participants affected / at risk) | 3/38 | 2/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | As Needed Dosing (N=38) | Continuous Infusion (N=40)
Severe adverse event (Cardiac disorders) | 0 (0) | 1 (1) — A subject developed hypotension and was withdrawn from the study. This subject had been receiving the infusion with morphine and midazolam. Blood pressure continued to decline over the next five hours before a myocardial arrest and re-intubation.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | As Needed Dosing (N=38) | Continuous Infusion (N=40)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1) — Hypotensive on morphine/midazolam for less than one hour. No bolus given. Bolus of fluid given when removed from study and blood pressure improved.
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Treating physician felt subject had a depressed respiratory drive. Subject had morphine/midazolam drip. No documentation of high carbon dioxide. Subject removed from study.
Paradoxical reaction to midazolam (Nervous system disorders) | 1 (1) | 0 (0) — On sixth dose of midazolam over an afternoon, subject was 'not acting himself'. Removed from study due to presumed paradoxical reaction
Inadequate pain control (Nervous system disorders) | 1 (1) | 0 (0) — Inadequate pain control per treating physician. Subject removed and dexmedetomidine started.
Large dose of acetaminophen given (Hepatobiliary disorders) | 1 (1) | 0 (0) — Inadvertent delivery of 60 mg/kg of acetaminophen instead of the 30 mg/kg in the protocol. Subject removed from study. No significant rise in ALT.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No